CLINICAL TRIAL: NCT00539565
Title: Phase IIIb Study of Corticosteroids as Post-Operative Adjuvant Therapy in Biliary Atresia
Brief Title: RCT of Steroids Following Kasai Portoenterostomy for Biliary Atresia.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: King's College Hospital NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCH99LG21
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-09

CONDITIONS: Biliary Atresia
Keywords: biliary atresia; Kasai portoenterostomy; corticosteroids
MeSH Terms: conditions — Biliary Atresia | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): oral corticosteroids
  Interventions: Drug: prednisolone
- B (Placebo Comparator): as for active regimen
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prednisolone — 2 mg/kg /day from post-op day 7 - day 21
  1 mg/kg /day from post-op day 22 - day 30
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
Biliary atresia is a congenital disorder of bile duct development or destruction of established but immature bile ducts. The study tests the hypothesis that post-operative steroids improve outcome following the Kasai procedure - the commonest surgical treatment.

DETAILED DESCRIPTION:
Biliary atresia is a potentially fatal condition of infants presenting as persisting jaundice in the first few weeks of life. The disease is characterised by obstruction and damage to the intra and extrahepatic parts of the biliary tree. Within the liver there is also a pronounced inflammatory response. The initial treatment is an attempt, by surgery, to restore bile flow by excising the obliterated extrahepatic bile ducts and joining part of the intestine to the bile "root" of the liver (the porta hepatis). This is known as the Kasai procedure. This is successful in ~50% of cases in reducing the level of jaundice to near-normal values. The use of steroids post-operatively has been suggested as improving outcome by diminishing the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* biliary atresia

Exclusion Criteria:

* <100 days at portoenterostomy
* no other anomalies (e.g. Biliary Atresia Splenic Malformation syndrome)
* anu contra-indications to corticosteroids

Max Age: 100 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
clearance of jaundice (<20 umol/L) | 1 year
Proportion transplanted or died | 1 year

SECONDARY OUTCOMES:
biochemical indices of liver function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark Davenport, ChM, Principal Investigator — Kings College Hospital
Locations (1):
- Kings College Hospital, London, United Kingdom